CLINICAL TRIAL: NCT01753947
Title: Individualized Deliberate Practice on a Virtual Reality Simulator Improves Technical Performance of Surgical Novices in the Operating Room: A Randomized Controlled Trial
Brief Title: Individualized Deliberate Practice on a Virtual Reality Simulator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Royal College of Physicians and Surgeons of Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: Deliberate Practice
Record Dates: First submitted 2012-12-07; First posted 2012-12-20 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2012-12

CONDITIONS: Education; General Surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Deliberate Practice (Experimental): Residents in the deliberate practice group received individualized feedback at the end of the initial assessment case. The staff surgeon supervising the case completed 3 previously validated technical skills assessment forms.
  Interventions: Other: Deliberate Practice
- Conventional Feedback (No Intervention): Residents in the control group received informal feedback as they performed the initial laparoscopic cholecystectomy in the operating room. This was left up to the discretion of the staff surgeon supervising the operation. This corresponds to the routine teaching and feedback practices that occur during conventional surgical residency training

INTERVENTIONS:
Other: Deliberate Practice
  Arms: Deliberate Practice

SUMMARY:
Training on simulated models in a surgical skills laboratory has been shown to improve technical performance in the operating room. Currently described simulation-based curricula consist of trainees practicing the same tasks until expert proficiency is reached. It has yet to be investigated whether individualized deliberate practice, where curricula tasks vary depending on prior levels of technical proficiency, would translate to the operating room.

This randomized controlled trial effectively demonstrates that deliberate practice on a virtual reality simulator results in an improvement in technical skills in a real clinical situation. This enhances the feasibility of implementing simulation-based curricula into residency training programs, and consequently has the potential to improve patient safety.

ELIGIBILITY:
Inclusion Criteria:

* post graduate year 1 and 2 surgical residents
* performed less than 10 laparoscopic cholecystectomies as the primary surgeon

Exclusion Criteria:

* n/a

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Technical skills | 6 months
  Participants' technical skills will be assessed in the operating room as they perform a laparoscopic cholecystectomy under supervision. The procedure will be video-recorded and sent for assessment to a blinded evaluator. Technical skills will be assessed using a previously validated technical skills assessment tool (Objective Structured Assessment of Technical Skill - OSATS)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Toronto, Toronto, Ontario, Canada